CLINICAL TRIAL: NCT05858866
Title: The Effects of Smartphone Addiction on Physical Activity, Fatigue and Sleep Quality of University Students
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tahir Keskin , Pt, MSc, Research Assistant, Suleyman Demirel University
Other Study IDs: SuleymanDUtahirkeskin02
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Addictive Behavior
MeSH Terms: conditions — Behavior, Addictive | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone-addicted group: university sdudents
  Interventions: Other: Piper Fatigue Scale
- non-smartphone-addicted group: university sdudents
  Interventions: Other: Piper Fatigue Scale

INTERVENTIONS:
Other: Piper Fatigue Scale — The Piper Fatigue Scale (PFS) was developed by Piper et al. to measure fatigue in a multi-dimensional manner. The scale assesses the behavioural, affective, sensory and cognitive/mood attributes of fatigue and contains 22 items and 5 open-ended questions. Each item is scored between 0 and 10 using a Visual Analogue Scale. Sub-scale scores are obtained by dividing the scores from the sub-scale items by the number of the items in the sub-scale. The same method is used to calculate the total score
  Other Names: Pittsburgh Sleep Quality Index; Physical Activity

SUMMARY:
The increasing rate of usage of smartphones ushers in various health problems and smartphone addiction. In the literature, the research focused mainly on the relationship between smartphone addiction and depression, anxiety and musculoskeletal system problems; however, the number of studies on fatigue was limited. We believe that this paper will be of interest to the readers of your journal because it adds information about the effect of smartphone addiction on physical activity, on sleep quality and especially on fatigue.

DETAILED DESCRIPTION:
This cross-sectional study was conducted with the participation of 322 students attending the Faculty of Health Sciences at Süleyman Demirel University. The participants were given the socio-demographic characteristics form, developed by the researchers according to the literature review. They were also given the evaluation form, which surveys some variables related to smartphones, as well as the short version of the Smartphone Addiction Scale Short Version (SAS-SV), the International Physical Activity Questionnaire-Short Form (IPAQ-SF), the Pittsburgh Sleep Quality Index (PSQI), and the Piper Fatigue Scale (PFS).

ELIGIBILITY:
Inclusion Criteria:

* The students who volunteered to participate in the study after being informed about the aims and procedures of the study.

Exclusion Criteria:

* The students who didnot volunteered to participate in the study after being informed about the aims and procedures of the study.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: University Students
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Short Version of the Smartphone Addiction Scale Short Version | 02.01.2021

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Merkez, Turkey (Türkiye)